CLINICAL TRIAL: NCT01192750
Title: Retrospective Analysis of ERCC1 Expression in Patients With Recurrent/Metastatic Squamous Cell Carcinoma of the Head and Neck (SCCHN) Who Received Cisplatin or Cisplatin and Cetuximab
Brief Title: Biomakers in Tissue Samples From Patients With Recurrent and/or Metastatic Squamous Cell Cancer of the Head and Neck Previously Treated With Cisplatin With or Without Cetuximab
Status: Completed | Type: Observational
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: CDR0000683281; ECOG-E5397T1
Record Dates: First submitted 2010-08-31; First posted 2010-09-01 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Head and Neck Cancer
Keywords: recurrent metastatic squamous neck cancer with occult primary; recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent verrucous carcinoma of the larynx; recurrent verrucous carcinoma of the oral cavity; stage IV verrucous carcinoma of the larynx; stage IV verrucous carcinoma of the oral cavity; recurrent salivary gland cancer; salivary gland squamous cell carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Salivary Gland Neoplasms | interventions — Immunohistochemistry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Other: medical chart review

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is studying biomarkers in tissue samples from patients with recurrent and/or metastatic squamous cell cancer of the head and neck previously treated with cisplatin with or without cetuximab.

DETAILED DESCRIPTION:
OBJECTIVES:

* To investigate the association between ERCC1 expression and clinical outcomes (response rate, progression-free survival, and overall survival) in patients with recurrent and/or metastatic squamous cell carcinoma of the head and neck who received cisplatin with versus without cetuximab on clinical trial ECOG-E5397.

OUTLINE: Archived tumor tissue samples are analyzed for ERCC1 expression by IHC. ERCC1 levels (low or high) are assessed by an H-score and AQUA, a quantitative IHC analysis. Each patient's ERCC1 level result is then compared with the patient's clinical outcome.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of squamous cell carcinoma of the head and neck

  * Recurrent and/or metastatic disease
* Received cisplatin with or without cetuximab on clinical trial ECOG-E5397
* Slides and blocks of tumor specimens available

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples from patients enrolled on E5397 from whom samples were submitted for research
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2010-08-05 (Actual); Primary Completion 2010-10-05 (Actual); Study Completion 2010-10-05 (Actual)

PRIMARY OUTCOMES:
Association between ERCC1 expression (low or high) with clinical outcomes | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Ranee Mehra, MD, Principal Investigator — Fox Chase Cancer Center